CLINICAL TRIAL: NCT02707419
Title: Self-administered Action Observation Treatment Enhance the Efficacy of Inpatient Rehabilitation After Total Knee Replacement: A Randomized Controlled Trial
Brief Title: Action Observation in Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dongnocchi
Record Dates: First submitted 2016-02-27; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Total Knee Replacement
Keywords: Total knee replacement; Action observation treatment; Rehabilitation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Video of the exercises and conventional physiotherapy. 45 minutes twice a day, 5 days a week for 2 weeks.
  Interventions: Device: Experimental group; Device: Conventional physiotherapy
- Control group (Active Comparator): Video of nature scenes and conventional physiotherapy. 45 minutes twice a day, 5 days a week for 2 weeks.
  Interventions: Device: Control group; Device: Conventional physiotherapy

INTERVENTIONS:
Device: Experimental group — Video of the exercises
  Arms: Experimental group
Device: Control group — video of nature scenes
  Arms: Control group
Device: Conventional physiotherapy — Mobilization, exercises and transfer practice.

SUMMARY:
Postoperative rehabilitation is required for a successful outcome following total knee arthroplasty. Traditionally rehabilitative programs aim to increase range of motion, to strengthen quadriceps, to restore normal gait, and to recover independence in activities of daily living. In the last decade action observation treatment, in addition to conventional physiotherapy has been proposed as a treatment method in rehabilitative medicine. There is growing evidence of the applicability of action observation training in rehabilitative medicine, indeed it has been applied in the rehabilitation of stroke of Parkinson disease of cerebral palsy and of aphasia.

Nevertheless those are small studies and one of them included a mixed population of hip and knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacement.

Exclusion Criteria:

* bilateral knee replacement
* previous total knee replacement.
* pre-existing motor impairment (i.e. hemiparesis, poliomyelitis, lumbar sciatica);

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity | Baseline and immediately post-intervention
  Visual Analogue Scale
Change of Range Of Motion | Baseline and immediately post-intervention
  Active and passive range of motion of knee

SECONDARY OUTCOMES:
Barthel index | Baseline and immediately post-intervention
  Barthel index
Short Form-36 motor | Baseline and immediately post-intervention
Tinetti scale | Baseline and immediately post-intervention
Lequesne index | Baseline and immediately post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Hugo Villafañe, Piossasco, Turin, Italy

IPD SHARING:
Plan to Share IPD: No